CLINICAL TRIAL: NCT06161480
Title: The Feasibility and Acceptability of Using Weighted Blankets to Prevent and/or Mitigate Delirium in Adult Critical Care Patients in Urban and Rural Settings.
Brief Title: Feasibility and Acceptability of Using Weighted Blankets to Prevent and /or Mitigate Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20027241
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Pilot study that will be conducted in a convenience sample of adult medicine ICU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Weighted Blanket (Other): To prevent and or mitigate delirium in adult ICU patients in urban and rural populations.
  Interventions: Device: Weighted Blanket

INTERVENTIONS:
Device: Weighted Blanket — Weighted Blanket is an occupational therapy modality which has been associated with significant increases in grounding, orientation to reality, soothing, and quality of life.

SUMMARY:
The use of weighted blankets to avert or alleviate Delirium in Adult ICU patients.

DETAILED DESCRIPTION:
To examine the feasibility and acceptability of weighted blankets as a single component, nonpharmacologic strategy to prevent and/or mitigate delirium in an adult medicine critical care patient population. To examine the feasibility and acceptability of videoconferencing (VCU Health Zoom), EHR screening, and VCU and VCU Health infrastructure (REDCap, OnCore) for rural participant recruitment and research participation, remote HealthCare provider protocol training and research engagement, and remote research monitoring and support for rural patient population. To collect preliminary descriptive data and examine trends related to the use of weighted blankets to prevent and/or mitigate delirium to inform future efficacy trials in an adult medicine critical care patient population (e.g., Agitation, Delirium, ICU length of stay, number ventilator days, sedation/opioid medication usage).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Requiring ICU level of care.
* Have a primary medical diagnosis.
* Proficient in English.

Exclusion Criteria:

* BMI less than 18.5.
* Significant deficit in cognitive functioning that is not expected to improve due to an end---stage disease stage or permanent injury (e.g., end-stage encephalopathy, traumatic or anoxic brain injury, dementia).
* Known pregnancy.
* Prisoners.
* Presence of skin injury (e.g., surgical wound, pressure injury, moisture injury) in an anatomical location where additional weight/pressure of blanket could prevent healing and /or lead to an expansion of the injury.
* Patients with skin injuries to areas easily left uncovered by the blanket (e.g., hands, feet) can be enrolled with additional communication to clinical team to leave areas uncovered to prevent additional injury.
* Paralysis effecting an area the weighted blanket will cover.
* Current neuromuscular blocking agent.
* Presence of recent/unhealed fractures on an area the blanket will cover (e.g., lower limb long bone, rib, pelvis, spine).
* History of claustrophobia reported by patient and/or their legally authorized representative (LAR).
* Fever of 37.5°C (99.5°F).
* Limited English proficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Study Participants Experience Survey | Six months
  Study Participants will be asked to complete a survey describing their experience with using the weighted blanket upon discharge from the ICU or if they stop using the weighted blanket, to determine if participants felt using the weighted blanket was beneficial to their overall health improvement.
LAR Experience Survey | Six Months
  LAR will complete survey describing his/her perspective of the participant's use of the weighted blanket to improve family member's health outcome. LAR will complete survey after participant has been discharged from ICU or participant is no longer using the weighted blanket.
Nurse and Provider Experience Survey | Six Months
  The nurse and healthcare provider will complete surveys once their patient has completed the use of the weighted blanket describing whether they felt the weighted blanket improved the health outcome of their patients.

SECONDARY OUTCOMES:
Analysis of total ICU Length of Stay (Days) | Six Months.
  Study Team will collect data daily and conduct analysis of total ICU Length of Stay (Days).
Analysis of total ICU Length of Stay on Study (Days) | Six Months
  Study Team will collect data daily and conduct analysis of total ICU Length of Stay on Study (Days)
Analysis of total Number of Ventilator Days (This admission) | Six Months
  Study Team will collect data daily and conduct analysis of total Number of Ventilator Days (This admission).
Analysis of total number of Ventilator Days on Study | Six Months
  Study Team will collect data daily and conduct analysis of total number of Ventilator Days on Study.
Daily Chart Review | Six Months
  Study Team will collect data daily and conduct analysis of the daily chart review data.
Blanket Usage Log analysis | Six Months
  Study Team will collect data daily and conduct analysis of the Blanket Usage Log.
Confusion Assessment Method for the ICU (CAM-ICU) data analysis | Six Months
  Study Team will collect data daily and conduct analysis of data from the CAM-ICU, a rating scale used be bedside clinicians to assess delirium for patients in the intensive care unit. The CAM-ICU-7 evaluates the presence of acute onset or fluctuating course (score of 0 or 1), inattention (score ranges from 0-2), altered level of consciousness (score ranges from 0-2, based on if RASS is anything other than alert and calm [zero]), and disorganized thinking (score ranges from 0-2).

CONTACTS AND LOCATIONS:
Locations (1):
- VCU Health Systems, Richmond, Virginia, United States